CLINICAL TRIAL: NCT06899867
Title: Is Cardiac Index, Assessed by Transpulmonary Thermodilution, Reliable During Liver Transplantation Compared to Transesophageal Echocardiography : a Monocentric Cohort
Brief Title: Comparing Montiroing Cardiac Index by Transpulmonary Thermodilution and Transesophageal Echocardiography During Liver Transplantation
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 24-5431
Record Dates: First submitted 2025-03-21; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Liver Transplantation
MeSH Terms: interventions — Thermodilution

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing liver transplantation at Croix-Rousse University Hospital, HCL, Lyon.: * Monitoring transesophageal echography, transpulmonary thermodilution
  * Measuring cardiac index, preload dependence (end-expiratory test) at 4 steps of surgery
  * Surgical anastomosis echography
  * Demographic data, biological data, post operation data
  Interventions: Other: Measure of cardiac index with thermodilution and transesophageal echocardiography; Other: Surgical anastomosis echography

INTERVENTIONS:
Other: Measure of cardiac index with thermodilution and transesophageal echocardiography — At 4 times of surgery, end-expiratory occlusion (EEO) test and measure of cardiac index before and after test with ETO and thermodilution
Other: Surgical anastomosis echography — Visualisation of surgical anastomosis through transesophageal echocardiography : stenosis, doppler velocity, collar diameter

SUMMARY:
Liver transplantation poses challenges due to hemodynamic changes throughout different surgical phases. Monitoring devices are essential for therapeutic adjustments. Transpulmonary thermodilution and transesophageal echocardiography are commonly used, but thermodilution may have limitations depending on the surgery.

This study aims to compare cardiac index variations between thermodilution and transesophageal echocardiography during liver transplantation. Patients undergo monitoring with both techniques. Measurements are recorded and reported at multiple time points.

ELIGIBILITY:
Inclusion Criteria:

* liver transplantation
* adults

Exclusion Criteria:

* - Oesophageal varice ligation < 14 days
* Mediastinal radiotherapy
* Femoral bypass
* Severe lower extremity artery disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: age > 18 years old, undergoing liver transplantation at Croix-Rousse hospital, HCL, Lyon
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac index variation measured by thermodilution compared with transesophageal echography | At 4 times of surgery: after starting anesthesia, anhepatic phase, reperfusion and surgical anastomosis of biliary ducts. Data reported : - Cardiac Index before and after end-expiratory test. - Transoesophageal echography measurement of cardiac function

CONTACTS AND LOCATIONS:
Locations (1):
- Croix Rousse Hsopital, France, Lyon, France